CLINICAL TRIAL: NCT06533813
Title: Clinical Epidemiology in Contemporary Patients With Myelofibrosis (ERNEST-3): A European LeukemiaNet (ELN) Observational Study
Brief Title: Clinical Epidemiology in Contemporary Patients With Myelofibrosis.
Acronym: ERNEST-3
Status: Recruiting | Type: Observational
Sponsor: FROM- Fondazione per la Ricerca Ospedale di Bergamo- ETS (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: ERNEST-3
Record Dates: First submitted 2024-07-19; First posted 2024-08-01 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Multicenter retrospective and prospective European observational study. At each site, all consecutive patients with a 2016- or 2022 World Health Organization (WHO) confirmed diagnosis of myelofibrosis (MF) established from 01/01/2018 to 31/12/2027 will be enrolled into the study. Yearly follow-up updates will be scheduled until the end of data collection on 31/12/2028 or until the last available patient visit, whichever comes first. At least 1 year of follow-up will be ensured from the last patient enrolled.

DETAILED DESCRIPTION:
Myeloproliferative neoplasms (MPNs) are rare bone marrow disorders characterized by clonal proliferation of hematopoietic cell lineages, and include polycythemia vera (PV), essential thrombocythemia (ET), and myelofibrosis (MF). MF has worse prognosis, with main causes of death including acute leukemia transformation, comorbid conditions, and consequences of cytopenia. MF is characterized by progressive anemia, bone marrow fibrosis, and extramedullary hematopoiesis with splenomegaly. Moreover, the disease is associated with a heavy symptom burden including night sweats, fever, bone pain, and weight loss and worsening the quality of life.

On the beginning of 2013 the European Registry for Myeloproliferative Neoplasms (ERNEST) observational study was launched and approved by several IRBs of European hematological centers. The study focused on overt Primary (PMF) and Secondary myelofibrosis (SMF; i.e., post-Essential Thrombocythemia myelofibrosis (post-ET MF) and post-polycythemia (post-PV MF)) and aimed at describing the clinical epidemiology of large series of patients observed in clinical practice. This research was justified as the landscape of both pathophysiological and clinical knowledge in MPNs was rapidly evolving, prompting to revise diagnostic criteria, prognostication and therapy recommendations.

ERNEST retrospectively enrolled 1292 patients in whom the proposed prognostic models were confirmed to differentiate treatments in clinical practice, while ERNEST-2 reported results on critical events observed in 1010 of these cases during a median follow-up period of 5.4 years.4,5 The two studies closed in December 2022.

In the last decade, new diagnostic and prognostic findings have been accumulated and the availability of new approved drugs, based on results of several new clinical trials, influenced the therapy decision making in the real-world clinical practice. Therefore, the continuation of observational studies in present ERNEST-3 on large multicenter case series of patients with MF is timely and might refine the results of clinical trials.

The purpose of this study observational retrospective/prospective study is to gain information on MF associated cytopenias that represent a significant challenge in the contemporary patients with MF. Currently, there are few agents aimed at treating cytopenic MF, including immunomodulatory drugs, hypomethylating agents, and JAK inhibitors such as momelotinib and pacritinib, and development of new agents specifically tailored to this patient population remains an unmet need. Therefore, this study can provide data on these patients, focusing on clinical status, quality of life, comorbidities, and treatment results over time.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary myelofibrosis (PMF) or secondary (i.e., post-ET/PV MF) myelofibrosis according to 2016- or 2022-WHO criteria ascertained between 01/01/2018 and 31/12/2027
* Age ≥ 18 years
* Signed informed consent where applicable, in line with current European General Data Protection Regulation (GDPR) directives

Exclusion Criteria:

* Diagnosis of early/prefibrotic primary myelofibrosis
* Concurrent participation to interventional clinical trials in MF

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a 2016- or 2022-WHO confirmed diagnosis of MF established from 01/01/2018 to 31/12/2027 will be enrolled into the study.
  Patients with primary and secondary to ET and PV myelofibrosis, annotated for genetic and histological features, in relation to the presence of baseline (i.e., at MF diagnosis) or treatment-related cytopenias (i.e., reduced count of blood cells manifesting as anemia, thrombocytopenia and/or neutropenia).
Sampling Method: Probability Sample
Enrollment: 617 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2025-12-19 (Actual); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival according to the presence of cytopenias at diagnosis | At diagnosis during the baseline
  Obtained by medical health records normally filled out in clinical practice

SECONDARY OUTCOMES:
Frequency and types of cytopenias | At baseline; 1 year follow-up.
  Obtained by medical health records normally filled out in clinical practice
Treatments response and duration (according to modified IWG-MRT and ELN 2013 criteria, overall and by presence of cytopenias | At baseline; 1 year follow-up.
  Obtained by medical health records normally filled out in clinical practice
Incidence of major CV events (thrombosis and bleeding), overall and by presence of cytopenias and treatments received | At baseline; 1 year follow-up.
  Obtained by medical health records normally filled out in clinical practice
Incidence of disease progressions (MF accelerated phase, MF blast phase/acute myeloid leukemia (AML)), overall and by presence of cytopenias and treatments received | At baseline; 1 year follow-up.
  Obtained by medical health records normally filled out in clinical practice
Incidence of secondary neoplasia, overall, by site and by presence of cytopenias and treatments received | At baseline; 1 year follow-up.
  Obtained by medical health records normally filled out in clinical practice
Incidence of infections, overall and by presence of cytopenias and treatments received | At baseline; 1 year follow-up.
  Obtained by medical health records normally filled out in clinical practice
Incidence of adverse events (AEs) of interest, overall, by type, severity and treatments received | At baseline; 1 year follow-up.
  Obtained by medical health records normally filled out in clinical practice
Incidence of death, overall, by cause and by presence of cytopenias and treatments received | At baseline; 1 year follow-up.
  Obtained by medical health records normally filled out in clinical practice

CONTACTS AND LOCATIONS:
Overall Officials: TIZIANO BARBUI, MD, Study Director — FROM- Fondazione per la Ricerca Ospedale di Bergamo- ETS
Locations (36):
- Hematology Center after Prof.R.H. Yeolyan, Yerevan, Armenia
- University of Copenhagen's Roskilde Hospital, Copenhagen, Denmark
- Clinical Investigation Center of the Saint Louis Hospital, Paris, France
- Germany (3):
  - Internal Medicine C, Hematology, Oncology, Stem Cell Transplantation and Palliative Care, University Medicine Greifswald, Greifswald
  - University Hospital Halle Department of Hematology/Oncology, Halle
  - University Clinic for Hematology, Oncology, Hemostaseology and Palliative Care Johannes Wesling Medical Center Minden UKRUB, University of Bochum, Minden
- Division of Haematology, Sasson University Hospital Assuta Ashdod, Ashdod, Ben-Gurion University of Negev, Ashdod, Israel
- Italy (20):
  - A.S.O. SS. Antonio e Biagio e C.Arrigo, SC Ematologia, Alessandria
  - ASST Papa Giovanni XXIII, SC Ematologia, Bergamo
  - Policlinico S. Orsola - Malpighi, Unità di Ematologia, Bologna
  - Azienda Ospedaliero - Universitaria "Policlinico Vittorio Emanuele" - PO Gaspare Rodolico, Dipartimento di ematologia con Trapianto di midollo Osseo, Catania
  - AOU Careggi di Firenze, Divisione di Ematologia, Florence
  - ASST Grande Ospedale Metropolitano Niguarda, Divisione di Ematologia, Milan
  - Fondazione IRCCS Ca' Granda - Ospedale Maggiore Policlinico, Ematologia, Milan
  - Ospedale San Raffaele, Unità Operativa di Ematologia e Trapianto Midollo Osseo, Milan
  - Fondazione IRCCS San Gerardo dei Tintori, Monza
  - Azienda Ospedaliera Universitaria Federico II, Divisione di Ematologia, Napoli
  - Azienda Ospedaliero Universitaria Maggiore della Carità, SCDU Ematologia, Novara
  - Azienda Ospedale-Università di Padova, Dipartimento di Medicina, Padua
  - Università degli Studi di Padova - Policlinico Universitario, Clinica Medica 1, Padua
  - Fondazione IRCCS Policlinico San Matteo, Divisione di Ematologia, Pavia
  - Fondazione Policlinico Universitario A. Gemelli - Università Cattolica del Sacro Cuore, UCSC Ematologia, Roma
  - Policlinico Umberto I, Dipartimento Ematologia, Oncologia e Dermatologia, Roma
  - A.O.U. Città della Salute e della Scienza di Torino - Ospedale Molinette- S.C. Ematologia U, Torino
  - ASST dei Sette Laghi (Ospedale di Circolo e F. Macchi), Divisione U.O. Ematologia, Varese
  - Azienda Ospedaliera Universitaria Integrata - Ospedale Borgo Roma, Unità di Ematologia, Verona
  - Azienda ULSS 8 Berica - Ospedale San Bortolo, Divisione di Ematologia, Vicenza
- Institute of Oncology, State University of Medicine and Pharmacy - Department of Oncology, Hematology and Radiotherapy, Chisinau, Moldova
- Poland (2):
  - Department of Hematology, University Hospital, Jagiellonian University Medical College, Krakow
  - Department and Clinic of Haematology, Blood Neoplasms, and Bone Marrow Transplantation, Wroclaw Medical University, Wroclaw
- Department of Hematology and Bone Marrow Transplantation, Fundeni Clinical Institute, Bucharest, Romania
- Spain (3):
  - Institut d'Investigacions Biomèdiques August Pi i Sunyer (IDIBAPS) - Hospital Clinic, Barcelona
  - Hematology and Hemotherapy Department, 12 de Octubre University Hospital, Madrid
  - Servicio de Hematología - Hospital Clínico Universitario de Valencia, Valencia
- United Kingdom (2):
  - School of Medicine, Dentistry and Biomedical Sciences Queen's University Belfast, Belfast
  - Guy's and St. Thomas' NHS Foundation Trust., London